CLINICAL TRIAL: NCT02859402
Title: Allogeneic Stem Cell Transplantation With 3-days Busulfan Plus Fludarabine as Conditioning in Patients With Relapsed or Refractory T-, NK/T-cell Lymphomas
Brief Title: Allogeneic Stem Cell Transplantation in Relapsed/Refractory T-, NK/T-cell Lymphomas
Acronym: RRTCLAlloSCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Young Rok Do, Prof., Keimyung University Dongsan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSMC 2016-05-051
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: T-cell Non-Hodgkin Lymphoma; Lymphoma, Extranodal NK-T-Cell
Keywords: T-cell Non-Hodgkin Lymphoma; NK/T-cell Non-Hodgkin Lymphoma; Relapsed, refractory; Conditioning; Allogeneic stem cell transplantation
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Extranodal NK-T-Cell; Recurrence | interventions — Busulfan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Arm (Experimental): Conditioning chemotherapy: Fludarabine and Busulfan followed by Allogeneic stem cell transplantation
  Interventions: Drug: Busulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Busulfan — intravenous, 3.2 mg/kg + 5% DW (the diluent quantity should be 10 times the volume of Busulfan, so that the final concentration of busulfan becomes approximately 0.5 mg/mL), once daily for 3 hours for 3 days (days -7 to -5)
  Other Names: Busulfex
Drug: Fludarabine — intravenous, 30 mg/m2 + 5% DW 100㎖, over 1 hour once daily for 6 days (days -8 to -3)

SUMMARY:
Relapsed and refractory T-cell lymphomas have been reported to have dismal outcomes. The role of allogeneic stem cell transplantation have been demonstrated in these patients. This clinical trial is studying the efficacy and safety of busulfan plus fludarabine as conditioning therapy followed by allogeneic stem cell transplantation (Allo-SCT) in T- and NK/T-cell lymphoma patients who have relapsed or are refractory to previous chemotherapies including autologous transplantation.

DETAILED DESCRIPTION:
Conditioning therapy

* Busulfan (Busulfex®; Patheon Manufacturing Services LLC, Greenville, NC 27834) 3.2 mg/kg + 5% DW (the diluent quantity should be 10 times the volume of Busulfan, so that the final concentration of busulfan becomes approximately 0.5 mg/mL), intravenously for 3 hours once daily for 3 days (days -7 to -5)
* Fludarabine (Fludarabine®, Zydus Hospira Oncology Private Ltd., Ahmedabad, India) 30 mg/m2 + 5% DW 100㎖, intravenously for over 1 hour once daily for 6 days (days -8 to -3)

  * Busulfan should be infused as soon as completion of fludarabine infusion

Primary objective of this study I. To determine the 2-year progression-free survival of this reduced toxicity conditioning in relapsed or refractory T- and NK/T-cell non-hodgkin lymphoma patients.

Secondary endpoints I. To evaluate the response rate, engraftment rate and time to engraftment, 2-year overall survival, 100-days treatment-related mortality, regimen-related toxicities by CTCAE version 4.03, post-transplantation complications (HVOD, acute/chronic graft-versus-host disease (GVHD), cytomegalovirus (CMV) infection,CMV disease) of this reduced toxicity conditioning in relapsed or refractory T- and NK/T-cell non-hodgkin lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 - 65
2. Histologically confirmed T or NK cell lymphomas :

   * anaplastic large cell lymphoma
   * angioimmunoblastic T-cell lymphoma,
   * peripheral T-cell lymphoma, NOS
   * NK/T-cell lymphoma
3. Relapsed after or refractory to one or more of previous chemotherapy including frontline autologous HSCT.
4. At least one measured lesion using conventional CT or PET CT at the time of relapse after or refractory to one or more of previous chemotherapy and before salvage chemotherapy
5. Complete or Partial response after short cycles of salvage chemotherapy
6. Patients who have HLA full-match (8/8 in HLA-A, B, C, DR by DNA high-resolution technique) or one-locus mismatch (7/8) sibling, or unrelated bone marrow or peripheral blood or cord blood stem cell donors
7. ECOG performance status ≤ 2
8. Charlson Comorbidity Index (CCI) before HSCT ≤ 3
9. Adequate renal function : serum creatinine level < 2.0 mg/dL
10. Adequate liver function :

    * Transaminase (AST/ALT) < 3 X upper normal value (or < 5 x ULN in the presence of lymphoma involvement of the liver)
    * Total bilirubin < 2 X upper normal value (or < 5 x ULN in the presence of NK/T involvement of the liver)
11. Cardiac ejection fraction ≥ 50 % as measured by MUGA or 2D ECHO without clinically significant abnormality
12. No clinically significant infection
13. No clinically significant bleeding symptoms or sign
14. Patients who decided to participate in this study and signed for a written consent

Exclusion Criteria:

1. Adult T cell leukemia/lymphoma, Lymphoblastic lymphoma, Primary cutaneous CD30+ T cell disorders Mycosis fungoides, Sezary SD
2. Patients who have previously performed Allo-HSCT
3. T cell lymphoma with primary central nervous system (CNS) Involvement.

   ** However, patients who have only had prophylactic intrathecal or intravenous chemotherapy against CNS disease are eligible.
4. Patients with a known history of HIV seropositivity or HCV (+).

   ** Patients with HBV are eligible. However, primary prophylaxis using antiviral agents is recommended for HBV carrier or prevent HBV reactivation during whole treatment period.
5. Any other malignancies within the past 5 years

   ** Except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
6. Ejection fraction < 50% by a echocardiography
7. FEV1 <60% or DLCO <60% by a pulmonary function test
8. ECOG performance status 3 or 4
9. Combined serious medical problem or disease

   * Serious or unstable heart disease although proper treatment
   * Myocardial infarction in recent 3 months
   * Underlying serious neurologic or psychiatric disease including dementia or seizure
   * Active uncontrolled infection including hepatitis B and C
   * Serious other medical problems observed by the doctors in charge of the patient
10. Pregnant or lactating women, women of childbearing potential not employing adequate contraception

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | 2 years
  2 year progression-free survival rate from the date of allogeneic stem cell transplantation. Estimated using the Kaplan-Meier method. Median value will be provided.

SECONDARY OUTCOMES:
Response rate | 3-months
  Response will be measured after 3 months of the date of allogeneic stem cell transplantation. Mean value will be provided.
Time to neutrophil engraftment | Day 30
  Summarized using standard descriptive statistics along with corresponding 95% confidence intervals.
Time to platelet engraftment | Day 30
  Summarized using standard descriptive statistics along with corresponding 95% confidence intervals.
2-year overall survival | 2 years
  2 year overall survival rate from the date of allogeneic stem cell transplantation. Estimated using the Kaplan-Meier method. Median value will be provided.
100-days treatment-related mortality | Days 100
  Summarized using standard descriptive statistics.
Rate of regimen-related toxicities | Day 30
  Toxicity according to CTCAE version 4.03. Summarized using standard descriptive statistics.
Rate of hepatic venoocclusive disease (HVOD) | Day 30
  Summarized using standard descriptive statistics.
Acute graft-versus-host disease (GVHD) grades I-IV | Day 100
  Summarized using standard descriptive statistics.
Chronic GVHD grades I-IV | 2 year
  Summarized using standard descriptive statistics.
Rate of cytomegalovirus (CMV) infection | 2 year
  Summarized using standard descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Dong-A University, Busan
  - Keimyung University Dongsan Medical Center, Daegu

IPD SHARING:
Plan to Share IPD: Yes
age,gender, disease type, stage, previous chemotherapy regimens, response to transplantation, patient survival, progression, toxicity profiles to the transpantation will be shared